CLINICAL TRIAL: NCT01611103
Title: Cognitive Effects of Transcranial Direct Current Stimulation in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Barry Gordon, M.D., Ph.D., Editor-in-Chief, Cognitive and Behavioral Neurology/Therapeutic Cognitive Neuroscience Professor/Professor of Neurology and Cognitive Science, Johns Hopkins University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 15657-O
Record Dates: First submitted 2012-05-31; First posted 2012-06-04 (Estimated); Last update posted 2015-09-01 (Estimated); Status verified 2015-08

CONDITIONS: Aging
Keywords: Cognitive Enhancement; tDCS; stimulation; elderly; older adults
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sham Stimulation (Sham Comparator): transcranial direct current stimulation that is ramped up and ramped down providing the sensation of tDCS without delivering the full amount of tDCS
  Interventions: Procedure: transcranial direct current stimulation
- Anodal Stimulation (Experimental): transcranial direct current stimulation using Anodal stimulation over the area of interest
  Interventions: Procedure: transcranial direct current stimulation

INTERVENTIONS:
Procedure: transcranial direct current stimulation — delivery of transcranial direct current stimulation or sham stimulation for 20 to 60 minutes

SUMMARY:
This research is being done to determine whether transcranial direct current stimulation (tDCS) can improve certain mental abilities. In this research, a 9 volt battery is used to deliver very weak electrical current to the surface of the scalp while participants complete cognitive tasks. Our aim is to find out whether tDCS will improve task performance in adults over the age of 55.

DETAILED DESCRIPTION:
Participants enrolled into this study may be asked to do the following:

* Grant permission for the researchers to view medical records associated with their language/cognitive difficulties (if applicable).
* Complete a questionnaire, provide a health history, and take some pencil-and-paper tests of problem-solving and memory in order to verify eligibility to participate and to able to safely undergo the experimental procedures.
* Complete several tasks (i.e., saying words out loud, naming objects, drawing designs, remembering lists of words, searching for images or letters, and/or completing puzzles) based upon a number of cognitive functions such as language, memory, vision, processing, and perception.
* Wear electrodes that will be placed on the scalp with a large rubberized band. These electrodes will administer very weak electrical current (tDCS) from a 9 volt battery for 20 to 60 minutes.
* Participate in several study conditions. The exact conditions and their order will be randomized. Under some conditions, participants may receive active stimulation (tDCS) and under other conditions, they may receive sham stimulation.
* The experimental sessions will last approximately 2 hours and participants may be asked to have more than one testing session in a day or to return for additional sessions.

ELIGIBILITY:
Inclusion Criteria:

* Over the age of 55
* Right Handed
* Native English speaker

Exclusion Criteria:

* History of Seizures
* Any implanted metal device or pacemaker
* Appreciable deficits in hearing or vision
* Greater than 1.5 standard deviations below demographically adjusted means on cognitive screen
* Dementia or Mini Mental Exam below 24

Ages: 55 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2012-06; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Cognitive Test Performance | The average time frame is 2 hours
  Cognitive test performance by subjects will be evaluated upon completion of enrollment to determine if tDCS improved performance on cognitive tests

CONTACTS AND LOCATIONS:
Overall Officials: Barry Gordon, Principal Investigator — Johns Hopkins University
Locations (1):
- Department of Neurology, Baltimore, Maryland, United States